CLINICAL TRIAL: NCT03252002
Title: Single/Multiple Dose Escalation Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BAY1101042 Given as 5 mg MR Tablet After Single Oral Dosing Followed by Once Daily Dosing for 7 Days in 12 Healthy Male Subjects Per Dose Step in a Randomized, Placebo Controlled, Single Blind, Group Comparison Design
Brief Title: Clinical Study to Evaluate the Pharmacokinetics, Safety, Tolerability and Pharmacodynamic Effects of a Single and Multiple Oral BAY1101042 Tablet Doses in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18747; 2017-001212-11 (EudraCT Number)
Record Dates: First submitted 2017-08-04; First posted 2017-08-16 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteer
Keywords: Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Single/multiple doses of 10 mg BAY1101042 or placebo (Experimental): Single oral dose of 10 mg BAY1101042 (given as 5 mg MR tablets) or corresponding placebo followed by once daily dosing for 7 days
  Interventions: Drug: BAY1101042; Drug: Placebo
- Single/ multiple doses of 20 mg BAY1101042 or placebo (Experimental): Single oral dose of 20 mg BAY1101042 (given as 5 mg MR tablets) or corresponding placebo followed by once daily dosing for 7 days
  Interventions: Drug: BAY1101042; Drug: Placebo
- Single/ multiple doses of 30 mg BAY1101042 or placebo (Experimental): Single oral dose of 30 mg BAY1101042 (given as 5 mg MR tablets) or corresponding placebo followed by once daily dosing for 7 days
  Interventions: Drug: BAY1101042; Drug: Placebo
- Single/ multiple doses of 40 mg BAY1101042 or placebo (Experimental): Single oral dose of 40 mg BAY1101042 (given as 5 mg MR tablets) or corresponding placebo followed by once daily dosing for 7 days
  Interventions: Drug: BAY1101042; Drug: Placebo
- Single/ multiple doses of 50 mg BAY1101042 or placebo (Experimental): Single oral dose of 50 mg BAY1101042 (given as 5 mg MR tablets) or corresponding placebo followed by once daily dosing for 7 days
  Interventions: Drug: BAY1101042; Drug: Placebo
- Optional: Single/multiple doses of 5 mg BAY 1101042 or placebo (Experimental): Single oral dose of 5 mg BAY1101042 MR tablets or corresponding placebo followed by once daily dosing for 7 days
  Interventions: Drug: BAY1101042; Drug: Placebo

INTERVENTIONS:
Drug: BAY1101042 — Single oral dose of 10 mg, 20 mg, 30 mg, 40 mg, 50 mg or optionally 5 mg BAY 1101042 (given as 5 mg MR tablets) or corresponding placebo followed by once daily dosing for 7 days
Drug: Placebo — Single dose on Day 1 (00d) and once daily for 7 days from Day 3 (02d) until Day 9 (08d)

SUMMARY:
To investigate the safety, tolerability, pharmacokinetics and effects of BAY1101042 in healthy male subjects after a single oral dose and multiple once daily dosing for 7 days

ELIGIBILITY:
Inclusion Criteria:

* The informed consent must be signed before any study specific tests or procedures are done.
* Healthy male subject.
* Age: 18 to 45 years (inclusive) at the screening.
* Body mass index (BMI): above/equal 18 and below/equal 29.9 kg/m2.
* Ability to understand and follow study-related instructions.

Exclusion Criteria:

* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal.
* Subjects with thyroid disorders as evidenced by assessment of thyroid stimulating hormone (TSH) levels outside the normal reference range at screening.
* Regular use of medicines.
* Smoking more than 10 cigarettes daily.
* Systolic blood pressure below 100 or above 145 mmHg (at screening).
* Diastolic blood pressure below 50 or above 90 mmHg (at screening).
* Heart rate below 50 or above 90 beats/ min (at screening).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | Approximately 19 days
  Assessment of treatment emergent adverse events from first study drug intake until follow up

SECONDARY OUTCOMES:
AUC(0-24) of BAY1101042 | At day 1
  AUC(0-24): area under the concentration vs. time curve from zero to 24 hours after single dose
AUC(0-24)/D of BAY1101042 | At day 1
  AUC(0-24)/D: dose-normalized area under the concentration vs. time curve from zero to 24 hours after single dose
Cmax of BAY1101042 | At day 1
  Cmax: maximum observed drug concentration after single dose
Cmax/D of BAY1101042 | At day 1
  Cmax/D: dose-normalized maximum observed drug concentration after single dose
AUCτ,md of BAY1101042 | At day 9
  AUCτ,md: area under the concentration vs. time curve for the actual dosing interval after multiple dose
AUCτ,md/D of BAY1101042 | At day 9
  AUCτ,md/D: dose-normalized area under the concentration vs. time curve for the actual dosing interval after multiple dose
Cmax,md of BAY1101042 | At day 9
  Cmax,md: maximum observed drug concentration after multiple dose
Cmax,md/D of BAY1101042 | At day 9
  Cmax,md/D: dose-normalized maximum observed drug concentration after multiple dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Germany (2):
  - CRS Clinical-Research-Services Mönchengladbach GmbH, Mönchengladbach, North Rhine-Westphalia
  - CRS Clinical Research Services Wuppertal GmbH, Wuppertal, North Rhine-Westphalia